CLINICAL TRIAL: NCT06510192
Title: Yuva Sath: A Peer-led Behavioral Intervention to Support Substance Use Treatment and HIV Prevention Among Young People Who Inject Drugs in India
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lakshmi Ganapathi, Physician-Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P000962; 1K23DA057151-01A1 (NIH)
Record Dates: First submitted 2024-07-04; First posted 2024-07-19 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Hiv; Substance Use Disorders
Keywords: Youth; India; People who inject drugs
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yuva Sath Intervention (Experimental): The Yuva Sath Intervention entails 6 one-on-one sessions delivered by peer counselors who will use an intervention manual consisting of modules and an intervention script. These sessions will occur over a period of 3 months. The intervention will also entail weekly check-in text messages from peer counselors. These weekly check-ins will occur over a period of 5 months.
  Interventions: Behavioral: Yuva Sath
- Treatment as usual (No Intervention): The treatment as usual arm consists of a single motivational interviewing session that will be provided by existing counselors at the integrated care center where the trial will take place. Participants in this arm will not receive the Yuva Sath Intervention

INTERVENTIONS:
Behavioral: Yuva Sath — The Yuva Sath Intervention comprises 6 one-on-one sessions with peer counselors who will use an intervention manual. The intervention also includes weekly phone text check-ins by peer counselors
  Arms: Yuva Sath Intervention

SUMMARY:
The goal of this pilot randomized controlled trial is to learn if Yuva Sath, a youth-tailored peer-led behavioral intervention, can support substance use treatment engagement and HIV prevention among young people who inject drugs in India. The main questions it aims to answer are:

* Is Yuva Sath feasible and is it acceptable to young people who inject drugs in India ?
* Can Yuva Sath improve engagement in substance use treatment, increase use of HIV prevention services and decrease substance use and risk behaviors among young people who inject drugs in India ?

Researchers will compare participants who receive the Yuva Sath behavioral intervention to participants who do not to see if the behavioral intervention improves substance use treatment engagement and HIV prevention.

Participants will:

* Receive a total of 6 one-on-one sessions, and weekly phone text check-ins from peer counselors over a course of 6 months.
* Complete monthly random urine drug screens
* Complete in-person study questionnaires every 3 months
* Report substance use and risk behaviors weekly to peer counselors through a brief phone text message survey

ELIGIBILITY:
Inclusion Criteria:

* Age 18-29 years;
* Receiving medications for opioid use disorder (MOUD) for at least 3 months and receipt frequency < 2 times a week

Exclusion Criteria:

* Receiving medications for opioid use disorder (MOUD) for less than 3 months and receipt frequency >= 2 times a week
* Requiring urgent medical attention
* Inability to provide informed consent

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Yuva Sath Intervention: Peer counselor fidelity | 6 months.
  Feasibility of the Yuva Sath intervention as measured by peer counselor fidelity to the intervention protocol will be determined by independent observer fidelity checklists. The checklist will score content delivery on a 3-point ordinal scale (1=no key content covered to 3=all key content covered), and peer-navigator actions (i.e., identification of barriers; generation of solutions) on a 5-point Likert scale (1=not at all to 5=very much). The intervention will be deemed to be feasible if 80% of the sessions addressed key Life-Steps module content and employed flexible problem-solving
Feasibility of the Yuva Sath Intervention: Attendance in the first four sessions | 6 months
  Feasibility of the Yuva Sath intervention as measured by attendance in the first four sessions will be calculated as a proportion: participants who completed the first four sessions of the total 6 sessions of the intervention/ All participants in the intervention arm. The intervention will be deemed to be feasible if at least 75% of participants completed the first four sessions
Feasibility of the Yuva Sath Intervention: Completion of the 3 month assessment | 3 months
  Feasibility of the Yuva Sath intervention as measured by completion of the 3 month session will be calculated as a proportion: participants who completed the 3 month assessment / All participants in the intervention arm. The intervention will be deemed feasible if at least 60% of participants completed the 3-month assessment
Acceptability of the Yuva Sath Intervention | 6 months
  Acceptability of the intervention as measured by the overall satisfaction of participants rated on a 5-point Likert scale (1=not at all to 5=very much). The intervention will be deemed acceptable if at least 75% of the participants rate >=4 on overall satisfaction

SECONDARY OUTCOMES:
Substance use treatment engagement: the number of MOUD visits each month | 6 months
  Substance use treatment engagement as measured by the average number of MOUD visits each month over a 6 month period will be compared between the intervention and control arms.
Substance use treatment engagement: the number of weeks of MOUD receipt at >2 times a week | 6 months
  Substance use treatment engagement as measured by the the number of weeks of MOUD receipt at >2 times a week will be compared between the intervention and control arms. We will calculate the proportion of participants (%) in each arm who on average received MOUD at a frequency of > 2 times a week.
Substance use treatment engagement: retention in MOUD at 6 months | 6 months
  Substance use treatment engagement as measured by retention in MOUD at 6 months will be compared between the intervention and control arms. We will calculate the proportion (%) of participants in each arm who were retained in MOUD at 6 months
HIV testing receipt | 6 months
  Receipt of regular HIV testing every 6 months will be compared between the intervention and control arms. We will calculate the proportion (%) of participants in each arm who received regular HIV testing
Substance use: Self report at 3-month assessment | 3 months
  Substance use as measured by self report will be compared between the intervention and control arms. We will calculate the proportion of participants (%) in the intervention and control arms who report continued substance use by at the 3-month assessment
Substance use: Self report at 6-month assessment | 6 months
  Substance use as measured by self report will be compared between the intervention and control arms. We will calculate the proportion (%) of participants in the intervention and control arms who report continued substance use by at the 6-month assessment
Substance use: monthly random point-of-care urinalysis | 6 months
  Substance use as measured by monthly point-of-care urinalysis will be compared between the intervention and control arms. We will calculate the proportion (%) of participants in the intervention and control arms who had at least one positive point-of-care test for opioids (excluding buprenorphine) in each arm
Needle sharing: Self report at 3-month assessment | 3 months
  Needle sharing as measured by self report will be compared between the intervention and control arms. We will calculate the proportion of participants (%) in the intervention and control arms who report needle sharing at the 3-month assessment
Needle sharing: self report at 6-month assessment | 6 months
  Needle sharing as measured by self report will be compared between the intervention and control arms. We will calculate the proportion of participants (%) in the intervention and control arms who report needle sharing at the 6-month assessment
Condomless sex: self report at 3-month assessment. | 3 months
  Condomless sex as measured by self report will be compared between the intervention and control arms. We will calculate the proportion of participants (%) in the intervention and control arms who report condomless sex at the 3-month assessment
Condomless sex: self report at 6-month assessment. | 6 months
  Condomless sex as measured by self report will be compared between the intervention and control arms. We will calculate the proportion of participants (%) in the intervention and control arms who report condomless sex at the 6-month assessment

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to other researchers at reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available once study analysis is completed and will be available for at least 5 years after study completion